CLINICAL TRIAL: NCT02367209
Title: Non-contrast-enhanced Perfusion Imaging of the Lung Using Fourier Decomposition Magnetic Resonance Imaging (FD MRI): Assessment of Feasibility in Patients With COPD in Correlation With Perfusion Scintigraphy, SPECT/CT and DCE MRI
Brief Title: Assessment of Lung Perfusion in Patients With Chronic Obstructive Pulmonary Disease Using FD MRI
Acronym: FD-COPD
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: FD-COPD-2015-002
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: COPD
Keywords: FD MRI; COPD; SPECT/CT; DCE MRI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In the recent years a novel method for functional lung imaging called Fourier decomposition MRI (FD MRI) has been introduced that allows for simultaneous assessment of regional lung perfusion and ventilation-related information without exposure to ionizing radiation or administration of intravenous or inhalational contrast agent. In this project, the investigators plan to investigate whether Fourier decomposition (FD) MRI is able to provide similar clinical information on regional lung perfusion as the standard methods SPECT/CT and DCE MRI in patients with COPD.

DETAILED DESCRIPTION:
In the recent years a novel method for functional lung imaging called Fourier decomposition MRI (FD MRI) has been introduced that allows for simultaneous assessment of regional lung perfusion and ventilation-related information without exposure to ionizing radiation or administration of intravenous or inhalational contrast agent.

In this project, the investigators plan to investigate whether Fourier decomposition (FD) MRI is able to provide similar clinical information on regional lung perfusion as the standard methods SPECT/CT and DCE MRI in patients with COPD. As MRI in patients with COPD is particularly challenging due to the rarefication of lung parenchyma, the FD MRI technique will be combined with an ultra-fast Steady-State Free Precession (ufSSFP) acquisition method for improved signal efficiency. The investigators ultimate goal is to provide a mean to predict and monitor the outcome of different therapies, such as medication, valves and surgery in COPD patients without requiring ionizing radiation or administration of contrast agents.

In the framework of this study, 30 patients with COPD will be enrolled prospectively. The study participants will be recruited by the clinic for thoracic surgery at the University Hospital Basel among all patients undergoing lung perfusion scintigraphy with SPECT/CT for surgery planning. Each participant will undergo one MRI examination of 30 min containing non-contrast-enhanced (FD MRI) and contrast-enhanced (DCE MRI) imaging studies of regional lung perfusion.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent as documented by signature

Exclusion Criteria:

* Known hypersensitivity or allergy to Gd-based MRI contrast agents.
* Patients with cardiac pacemakers, intra cranial clips, metallic foreign bodies^or other not MRcompatible implants (e.g. pumps etc.).
* Renal failure or severely impaired kidney function (eGFR < 30 ml/min /1,73 m2)
* Known or suspected non-compliance, claustrophobia.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Epilepsy.
* Age <18 years.
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study participants will be recruited by the department of thoracic surgery at the University Hospital Basel among all patients who undergo Perfusion scintigraphy and SPECT/CT of the lung with 99mTc-MAA for one of the following clinical indications (of note: this selection of patients does per se exclude pregnant women):
  1. Preoperative assessment of regional lung perfusion before video-assisted lung volume resection (VATS-LVRS) in patients with COPD.
  2. Preoperative assessment of regional lung perfusion before segmentectomy, lobectomy or pneumonectomy procedures with curative intention in NSCLC patients with concomitant COPD and reduced pulmonary function parameters (FEV1 < 80%).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Relative perfusion | 14 month
  Relative perfusion of individual pulmonary lobes expressed in % of total (bilateral) lung perfusion

SECONDARY OUTCOMES:
Image quality | 14 month
  Subjective classification by two independent readers
Perfusion defects | 14 month
  Inter-reader agreement concerning the presence of circumscribed perfusion defects

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bremerich, Prof., Principal Investigator — Klinik für Radiologie und Nuklearmedizin, Universitätsspital Basel
Locations (1):
- University of Basel Hospital, Clinic of Radiology and Nuclear Medicine, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No